CLINICAL TRIAL: NCT07340385
Title: The Effects of Training History on Physiological and Biochemical Responses in Blood Flow Restriction Strength Training
Brief Title: Physiological and Biochemical Responses to Blood Flow Restriction Training
Status: Not yet recruiting | Type: Observational
Sponsor: Afyonkarahisar Health Sciences University (Other)
Collaborators: Kocatepe University (Other)
Responsible Party: Principal Investigator, Fatma Eken, Research Assistant, Afyonkarahisar Health Sciences University
Other Study IDs: 2025/9
Record Dates: First submitted 2026-01-06; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Healthy Individuals; Trained Athletes
Keywords: Strength Training; Oxidative Stress; Growth Factors; Biochemical Markers; Muscle Thickness
MeSH Terms: interventions — Blood Flow Restriction Therapy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Novice Training Group: This group consists of healthy individuals who are new to strength training. Participants in this group will perform low-intensity resistance exercises with blood flow restriction applied to the proximal thigh using an inflatable cuff.
  Interventions: Other: Blood Flow Restriction Training
- Experienced Athletes Group: This group includes healthy experienced athletes from different sports disciplines and training load levels. Participants will perform the same low-intensity blood flow restriction exercise protocol applied to the proximal thigh using an inflatable cuff.
  Interventions: Other: Blood Flow Restriction Training

INTERVENTIONS:
Other: Blood Flow Restriction Training — Adaptation to blood flow restriction exercise training and the individually tailored occlusion pressure will be determined during the initial sessions. Occlusion pressure will be assessed while the participant is in a supine position by inflating a pneumatic cuff placed on the thigh until the tibial artery pulse is no longer detectable, which will be confirmed using a handheld Doppler device. To ensure safe adaptation to the training protocol, the pressure applied during the first two training sessions will be set below the individually determined target pressure. The full target occlusion pressure will be implemented starting from the third training session. For example, if the target pressure is determined as 300 mmHg, exercises will be performed at 200 mmHg during the first session and 250 mmHg during the second session. Blood flow restriction training principles will be applied during exercise loading. Four different types of exercises will be set up in four sets.

SUMMARY:
This study is designed to examine the short-term and long-term effects of blood flow restriction exercise training on physiological and biochemical markers in individuals who are new to strength training and in experienced athletes training at different load levels. This exercise method involves placing a special inflatable cuff around the upper part of the thigh. The cuff partially limits blood flow to the area, which helps the muscles work more effectively during exercise. The cuff will be applied only to the individual's dominant leg (the leg you use more often in daily activities), but all exercises will be performed using both legs. The exercise program will last for a total of six weeks and will be carried out twice per week. The pressure applied by the cuff will be individually adjusted based on each participant's physical characteristics to ensure safety and comfort. The study will include a total of 30 healthy participants aged between 18 and 40 years. Participants will be divided into two groups: individuals who have recently started strength training and experienced athletes with different levels of training experience.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation of healthy adults (both female and male)
* Age between 18 and 40 years
* No history of orthopedic pathology or current symptoms affecting the lower extremities
* For individuals with prior training experience: engagement in strength training at least two days per week for the past year across different sports disciplines
* For individuals new to strength training: no regular participation in strength training within the past six months

Exclusion Criteria:

* History of hypertension, cardiovascular diseases, peripheral vascular diseases, deep vein thrombosis, neurological disorders, obesity, or a diagnosis of diabetes
* Current or previous diagnosis of cancer
* Pregnancy
* Individuals who do not consent to participate in the study

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population consists of healthy adults aged 18-40 years, including individuals who are new to strength training and experienced athletes from different sports disciplines with varying training load levels.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2026-01-20 (Estimated); Primary Completion 2027-01-20 (Estimated); Study Completion 2027-03-20 (Estimated)

PRIMARY OUTCOMES:
Muscle Thickness | Baseline and after 6 weeks of training
Blood Biomarkers | Blood samples will be collected at three time points: before and immediately after the third training session to assess acute responses, and at the end of the 6-week training period to assess long-term effects.
  Oxidative Stress Markers Growth Factor Levels Muscle Damage Markers

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Nielsen JL, Aagaard P, Prokhorova TA, Nygaard T, Bech RD, Suetta C, Frandsen U. Blood flow restricted training leads to myocellular macrophage infiltration and upregulation of heat shock proteins, but no apparent muscle damage. J Physiol. 2017 Jul 15;595(14):4857-4873. doi: 10.1113/JP273907. Epub 2017 Jun 23. PMID 28481416
- [Result] Centner C, Zdzieblik D, Dressler P, Fink B, Gollhofer A, Konig D. Acute effects of blood flow restriction on exercise-induced free radical production in young and healthy subjects. Free Radic Res. 2018 Apr;52(4):446-454. doi: 10.1080/10715762.2018.1440293. Epub 2018 Mar 15. PMID 29448855
- [Result] Bernard J. [Complete remissions and current treatment of acute leukemia]. Probl Gematol Pereliv Krovi. 1965 Nov;10(11):3-9. No abstract available. Russian. PMID 5873262